CLINICAL TRIAL: NCT02629419
Title: A Phase 2a Efficacy, Safety, Tolerability, and PK Study of Encochleated Amphotericin B (CAMB/MAT2203) in Patients With Mucocutaneous Candidiasis Who Are Refractory or Intolerant to Standard Non-Intravenous Therapies
Brief Title: CAMB/MAT2203 in Patients With Mucocutaneous Candidiasis
Acronym: CAMB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Matinas BioPharma Nanotechnologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MB-70004; 16-I-0002 (Other: NIAID)
Record Dates: First submitted 2015-11-16; First posted 2015-12-14 (Estimated); Results first posted 2024-06-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-07

CONDITIONS: Candidiasis, Chronic Mucocutaneous
Keywords: STAT3 deficient Hyper IgE syndrome; Gain of function STAT1 defects; Autoimmune polyendocrinopathy-candidiasis-ectodermal dystrophy (APECED); IL-17/IL-22 autoantibodies from thymoma; Job's Syndrome (Hyperimmunoglobulin E Syndrome, Buckley Syndrome)
MeSH Terms: conditions — Candidiasis, Chronic Mucocutaneous; Polyendocrinopathies, Autoimmune; Job Syndrome | interventions — Amphotericin B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CAMB (Encochleated Amphotericin B) (Experimental): Encochleated Amphotericin B (200 mg, 400 mg, 800 mg)
  Interventions: Drug: Amphotericin B

INTERVENTIONS:
Drug: Amphotericin B — Oral lipid nanocrystal formulation of amphotericin B
  Other Names: Encochleated Amphotericin B; CAMB; MAT2203

SUMMARY:
This is an open-label, dose-titration trial to study the efficacy, safety, and pharmacokinetics of oral cochleate amphotericin B (CAMB) in the treatment of mucocutaneous candidiasis infections in patients who are refractory or intolerant to standard non intravenous therapies.

DETAILED DESCRIPTION:
Patients aged 18 to 75 years with mucocutaneous candidiasis (esophageal, oropharyngeal, or vulvovaginal) who are refractory or intolerant to standard non-intravenous therapies will be enrolled. Patients will initially be treated in a short-term dose titration period, where the dose may be increased in patients that do not respond clinically. Patients who do not respond clinically to the highest dose of drug will discontinue the protocol. Patients that respond to treatment and tolerate the study medication will be eligible to enter a long-term extension (up to 60-months).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a clinical diagnosis of at least one of the following:
* Persistent oropharyngeal candidiasis (OPC) for greater than or equal to 5 days documented on at least one occasion by potassium hydroxide (KOH) test or fungal stain and confirmed by mycological culture to be azole resistant within the previous 6 months and/or intolerance to standard non intravenous therapies or lack of improvement or worsening of OPC after receipt of appropriately dosed oral azole therapy.
* Esophageal candidiasis (EC) associated with clinical symptoms of retrosternal pain, odynophagia, and/or pain with swallowing and documented by esophageal biopsy or visualization with culture documenting azole resistance within the previous 6 months and/or intolerance to standard non-intravenous therapies or lack of improvement or worsening of EC after appropriately dosed azole therapy.
* Persistent vulvovaginal candidiasis (VVC) for greater than or equal to 5 days as documented by presence of vaginal symptoms and a positive wet mount showing Candida structures and confirmed by a vaginal culture positive for Candida with azole resistance within the previous 6 months and/or intolerance to standard non intravenous therapies or lack of improvement or worsening of VVC after appropriately dosed azole therapy.
* Patient is expected to survive for greater than or equal to 6 months.
* Willing to have samples stored for future research.
* Agree to use highly effective contraception.

  * Contraception: Because the effects of CAMB on the developing human fetus are unknown, sexually active patients of childbearing potential must agree to use highly effective contraception as outlined below before study entry and for the duration of study participation. Females of childbearing potential must have a negative pregnancy test result before receiving CAMB. During the course of the study, if a patient becomes pregnant or suspects they are pregnant, then they should inform the study staff and their primary care physician immediately. Acceptable forms of contraception are:

    * Intrauterine device (IUD) or equivalent.
    * Hormonal contraceptives (eg, consistent, timely and continuous use of contraceptive pill, patch, ring, implant, or injection that has reached full efficacy prior to dosing). If the patient uses contraceptive pill, patch, or ring, then a barrier method (eg, male/female condom, cap, or diaphragm plus spermicide) must also be used at the time of potentially reproductive sexual activity.
    * Be in a stable, long-term monogamous relationship, per principal investigator (PI) assessment, with a partner that does not pose any potential pregnancy risk, eg, has undergone a vasectomy at least 6 months prior to first dose of study agent or is of the same sex as the patient.
    * Have had a hysterectomy and/or a bilateral tubal ligation or both ovaries removed.

Exclusion Criteria:

* Allergy to any amphotericin B (AMB) product or any component of CAMB (eg, phosphatidylserine)
* Have evidence of systemic fungal infections requiring intravenous antifungal therapy
* Pregnant or nursing women, and women intending to become pregnant during the study period
* Had a concomitant medical condition that could interfere with study drug evaluation or that is a contraindication to the proposed investigational treatment based upon known agent safety profile or toxicities.
* Had any of the following laboratory abnormalities at the screening visit:

  * Alanine Transaminase (ALT), Aspartate Transaminase (AST) and Alkaline phosphatase (ALP) > 2.5 times the upper limit of normal (ULN).
  * Total bilirubin level > 2.5 times the ULN
  * Serum creatinine level > 2 times the ULN
  * Absolute neutrophil count less than 500 cells/microliter
  * Potassium level less than 3.5 mmol/L
* Exposure to any investigational agent within 4 weeks prior to Day 0 (Baseline).
* Current or recent history (past 12 months) of drug or alcohol abuse.
* Use of intravenous AMB products within 1-week of start of study drug administration
* Use of non-intravenous AMB products (such as oral AMB swishes) within 72 hours prior to start of study drug administration
* Any other condition the investigator believes would interfere with the patient s ability to provide informed consent, comply with study instructions, or which might confound the interpretation of the study results or put the subject at undue risk.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-09-27 (Actual); Primary Completion 2021-11-09 (Actual); Study Completion 2022-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Freeman, MD, Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institute of Allergy and Infectious Disease (NIAID), Bethesda, Maryland, United States

REFERENCES:
- [Derived] Desai JV, Urban A, Swaim DZ, Colton B, Kibathi LW, Ferre EMN, Stratton P, Merideth MA, Hunsberger S, Matkovits T, Mannino R, Holland SM, Tramont E, Lionakis MS, Freeman AF. Efficacy of Cochleated Amphotericin B in Mouse and Human Mucocutaneous Candidiasis. Antimicrob Agents Chemother. 2022 Jul 19;66(7):e0030822. doi: 10.1128/aac.00308-22. Epub 2022 Jun 14. PMID 35699443

RESULTS

PARTICIPANT FLOW:
Groups:
- MAT2203 (Previously Referred to as Encochleated Oral Amphotericin B [CAMB]): MAT2203 (200 mg, 400 mg, 800 mg)
  Oral lipid nanocrystal formulation of amphotericin B
Period: Overall Study
Arm/Group | MAT2203 (Previously Referred to as Encochleated Oral Amphotericin B [CAMB])
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | MAT2203 (Previously Referred to as Encochleated Oral Amphotericin B [CAMB])
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4
Chronic Mucocutaneous Candidiasis (CMC) Infection Type [Number; unit: participants]
  Oropharyngeal candidiasis (OPC) | 3
  Esophageal candidiasis (EC) | 1
  Vulvovaginal candidiasis (VVC) | 1

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response to Treatment of Mucocutaneous Candidiasis
Description: Number of subjects with a clinical response of clinical cure or improvement. Clinical cure was defined as absence of signs or symptoms of infection.
  Clinical improvement was defined as follows:
  * OPC or EC: partial resolution defined as greater than or equal to 50% of Baseline signs or symptoms
  * VVC: reduction of greater than or equal to 50% of clinical severity score from Baseline Severity of each symptom was graded on a scale from zero (absence of symptoms) to 3 (severe symptoms). The sum of all scores for all symptoms was used as the clinical severity score. Higher scores mean worse outcomes.
Time Frame: 14-days at highest titrated dose
Measure: Count of Participants; unit: Participants
Arm/Group | MAT2203 (Previously Referred to as Encochleated Oral Amphotericin B [CAMB])
Number analyzed (Participants) | 4
Participants | 4

2. Secondary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to 24 Hours Postdose
Description: Drug concentration in plasma collected at 0, 1, 2, 4, 8, 10, 12, and 24 hours post-dose
Time Frame: Single and Multiple Doses (14-days)
Population: 2 participants were not included in the analysis
Measure: Median (Inter-Quartile Range); unit: ng x h/mL
Arm/Group | MAT2203 (Previously Referred to as Encochleated Oral Amphotericin B [CAMB])
Number analyzed (Participants) | 2
ng x h/mL | 606 [435.18 to 777.17]

3. Secondary Outcome: Maximum Plasma Concentration (Cmax)
Description: Plasma concentration was measured at 0, 1, 2, 4, 8, 10, 12, and 24 hours post-dose
Time Frame: Single and Multiple Doses (14-days)
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | MAT2203 (Previously Referred to as Encochleated Oral Amphotericin B [CAMB])
Number analyzed (Participants) | 4
ng/mL | 28.4 [27.02 to 52.60]

4. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax)
Description: Plasma collected at 0, 1, 2, 4, 8, 10, 12, and 24 hours post-dose
Time Frame: Single and Multiple Doses (14-days)
Measure: Median (Inter-Quartile Range); unit: h
Arm/Group | MAT2203 (Previously Referred to as Encochleated Oral Amphotericin B [CAMB])
Number analyzed (Participants) | 4
h | 16 [4 to 24]

5. Secondary Outcome: Long-term Adverse Events, Changes in Laboratory Parameters
Description: Incidence of nephrotoxicity, defined as an increase of greater than 100% of baseline serum creatinine.
  Incidence of hypokalemia, defined as serum potassium less than or equal to 3mmol/L during or within 3 weeks of completing treatment.
Time Frame: up to 60 months
Measure: Number; unit: events
Arm/Group | MAT2203 (Previously Referred to as Encochleated Oral Amphotericin B [CAMB])
Number analyzed (Participants) | 4
events | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the entire study period up to 60 months
Description: Adverse events were noted at each study visit
Arm/Group | MAT2203 (Previously Referred to as Encochleated Oral Amphotericin B [CAMB])
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 3/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MAT2203 (Previously Referred to as Encochleated Oral Amphotericin B [CAMB]) (N=4)
Colostomy closure (Surgical and medical procedures) | 1
Pneumonia (Infections and infestations) | 2
Influenza (General disorders) | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Oral candidiasis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Subcutaneous abscess (Infections and infestations) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MAT2203 (Previously Referred to as Encochleated Oral Amphotericin B [CAMB]) (N=4)
Neutropenia (Blood and lymphatic system disorders) | 1
Tinnutis (Ear and labyrinth disorders) | 2
Vertigo (Ear and labyrinth disorders) | 1
Keratitus (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Hiatus Hernia (General disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Oesophageal ulcer (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 1
Chills (General disorders) | 1
Fatigue (General disorders) | 3
Malaise (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 2
Acute sinusitis (Infections and infestations) | 1
Clostridium defficile infection (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 1
Laryngitis (Infections and infestations) | 1
Mucocutaneous candidiasis (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Vulvitis (Infections and infestations) | 1
Vulvovaginal candidiasis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Fracture (Injury, poisoning and procedural complications) | 2
Injury (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Blood albumin decreased (Investigations) | 1
Blood bicarbonate abnormal (Investigations) | 1
Blood bicarbonate decreased (Investigations) | 1
Blood cholesterol increased (Investigations) | 1
Blood immunoglobulin E increased (Investigations) | 1
Blood immunoglobulin G increased (Investigations) | 1
Blood iron decreased (Investigations) | 2
Blood lactate dehydrogenase (Investigations) | 1
Blood potassium decreased (Investigations) | 1
Blood thyroid stimulating hormone increased (Investigations) | 1
Body temperature increased (Investigations) | 1
C-reactive protein increased (Investigations) | 3
Haemoglobin decreased (Investigations) | 2
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 1
Oxygen saturation abnnormal (Investigations) | 1
White blood cell count increased (Investigations) | 3
Decreased appetite (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 4
Hypernatraemia (Metabolism and nutrition disorders) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Musculoskelatal chest pain (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Aegusia (Nervous system disorders) | 1
Cognitive disorder (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 3
Tremor (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Bladder irritation (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 2
Vaginal discharge (Reproductive system and breast disorders) | 1
Vulvovaginal pruritis (Reproductive system and breast disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 3
Skin lesion (Skin and subcutaneous tissue disorders) | 3
Tooth extraction (Surgical and medical procedures) | 1
Haematoma (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Did not reach target number of participants (small sample size). All participants were female and Caucasian.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-01): https://cdn.clinicaltrials.gov/large-docs/19/NCT02629419/Prot_SAP_001.pdf
  • Informed Consent Form (2021-03-29): https://cdn.clinicaltrials.gov/large-docs/19/NCT02629419/ICF_000.pdf